CLINICAL TRIAL: NCT02753881
Title: Pharmacokinetics of Doxorubicin in Conventional Transarterial Chemoembolization (cTACE) of Primary and Secondary Liver Cancer
Brief Title: Pharmacokinetics of Doxorubicin in cTACE of Liver Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1506016008
Record Dates: First submitted 2016-03-10; First posted 2016-04-28 (Estimated); Results first posted 2020-08-03 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- whole liver lobe cTACE doxorubicin (Active Comparator): Participants in this arm are administered 10 cc of chemotherapy, with 50mg doxorubicin and 10 mg of mitomycin-C via cTACE delivered in a lobar (whole liver) manner.
  Interventions: Drug: whole liver lobe cTACE doxorubicin
- superselective cTACE doxorubicin (Active Comparator): Participants in this arm are administered 10 cc of chemotherapy, with 50mg doxorubicin and 10 mg of mitomycin-C via cTACE delivered in a super-selective (close to the tumor) manner.
  Interventions: Drug: superselective cTACE doxorubicin

INTERVENTIONS:
Drug: whole liver lobe cTACE doxorubicin — Doxorubicin CTACE administered in a whole liver lobe manner.
  Arms: whole liver lobe cTACE doxorubicin
Drug: superselective cTACE doxorubicin — Doxorubicin CTACE administered in a super-selective (close to the tumor) manner.
  Arms: superselective cTACE doxorubicin

SUMMARY:
Patients with primary and secondary liver cancer may participate in this study. The purpose is to perform an analysis of the effects of doxorubicin and its metabolite doxorubicinol on the body (doxorubicin pharmacokinetics ) after conventional transarterial chemoembolization (cTACE). cTACE is a procedure in which chemotherapy drugs are injected, followed by an injection of small beads to block the tumor-feeding arteries. Doxorubicin is a chemotherapeutic agent used in the cTACE procedure. This study will examine doxorubicin pharmacokinetics in patients who: 1) receive whole liver cTACE; and 2) receive super-selective CTACE (i.e., delivered in close proximity to the tumor).

DETAILED DESCRIPTION:
Patients with primary and secondary liver cancer may participate in this study. The purpose is to perform an analysis of the effects of doxorubicin and its metabolite doxorubicinol on the body (doxorubicin pharmacokinetics ) after conventional transarterial chemoembolization (cTACE). A pharmacokinetics profile (PK profile) will be constructed and will include peak of plasma concentration (Cmax), time of maximum concentration (TMax), and area under the concentration curve (AUC). This composite measure will be used to compare patients in cTACE lobar administration and cTACE superselective administration. In addition, the PK profile will be correlated with toxicity, tumor burden, body surface area, and gender. Feasibility and safety will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Histologically, cytologically, or radiologically confirmed liver dominant or liver only malignancy.
3. Preserved liver function (Child-Pugh A-B class) without significant liver decompensation.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 at study entry.
5. Measurable or evaluable disease that will be directly treated with intrahepatic therapy (as defined by Response Evaluation Criteria in Solid Tumors [RECIST] 1.1).
6. Suitable for TACE based on blood parameters such as platelet count, bilirubin, and international normalized ratio.
7. May be enrolled with a history of prior liver directed intra-arterial therapy if intra-arterial therapy to the target lesion occured > 1 year prior to enrollment date. Intra-arterial therapy to different targets within 1 year prior to enrollment date will not exclude subjects.

Exclusion Criteria:

1. Serum total bilirubin > 3.0 mg/dL
2. Creatinine > 2.0 mg/dL
3. Platelets < 50000/µL
4. Complete portal vein thrombosis with reversal of flow
5. Ascites (trace ascites on imaging is acceptable)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Schlachter, M.D., Principal Investigator — Yale University
Locations (1):
- Yale University, Department of Diagnostic Radiology, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Savic LJ, Chapiro J, Funai E, Bousabarah K, Schobert IT, Isufi E, Geschwind JH, Stark S, He P, Rudek MA, Perez Lozada JC, Ayyagari R, Pollak J, Schlachter T. Prospective study of Lipiodol distribution as an imaging marker for doxorubicin pharmacokinetics during conventional transarterial chemoembolization of liver malignancies. Eur Radiol. 2021 May;31(5):3002-3014. doi: 10.1007/s00330-020-07380-w. Epub 2020 Oct 15. PMID 33063185

RESULTS

PARTICIPANT FLOW:
Groups:
- Superselective cTACE Doxorubicin (One Segment): Participants in this arm are administered 10 cc of chemotherapy, with 50mg doxorubicin and 10 mg of mitomycin-C via Lipiodol cTACE delivered in a super-selective (close to the tumor) manner.
  superselective cTACE doxorubicin: Doxorubicin CTACE administered in a super-selective (close to the tumor) manner. Lipiodol delivered to single segment.
- Superselective cTACE (2+ Segments): Participants in this arm are administered 10 cc of chemotherapy, with 50mg doxorubicin and 10 mg of mitomycin-C via Lipiodol cTACE delivered in a super-selective (close to the tumor) manner.
  superselective cTACE doxorubicin: Doxorubicin CTACE administered in a super-selective (close to the tumor) manner. Lipiodol distributed to multiple segments.
- Whole Liver Lobe cTACE Doxorubicin: Participants in this arm are administered 10 cc of chemotherapy, with 50mg doxorubicin and 10 mg of mitomycin-C via Lipiodol cTACE delivered in a lobar (whole liver) manner.
  whole liver lobe cTACE doxorubicin: Doxorubicin CTACE administered in a whole liver lobe manner. Lipiodol distributed to entire liver lobe.
Period: Overall Study
Arm/Group | Superselective cTACE Doxorubicin (One Segment) | Superselective cTACE (2+ Segments) | Whole Liver Lobe cTACE Doxorubicin
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Superselective cTACE Doxorubicin (One Segment) | Superselective cTACE (2+ Segments) | Whole Liver Lobe cTACE Doxorubicin | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 8 | 17
  >=65 years | 4 | 7 | 2 | 13
Age, Continuous [Mean (Full Range); unit: years] | 63.7 [52 to 86] | 66.8 [54 to 76] | 59.1 [46 to 67] | 63.2 [46 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 3 | 5
  Male | 9 | 9 | 7 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 7 | 8 | 7 | 22
  More than one race | 1 | 1 | 1 | 3
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics Profile-- Peak of Plasma Concentration (Dose-normalized)
Description: Peak of plasma concentration (Cmax) of both doxorubicin and doxorubicinol reported for 10 lobar subjects, 10 superselective subjects with Lipiodol distribution to 1 segment, and 10 superselective subjects with Lipiodol distribution to multiple segments after dose normalization.
Time Frame: 0, 5, 10, 20, 40 minutes, 1, 2, 4, 24 hours, and 3-4 weeks post dose
Population: 6 of 10 lobar, 7 of 10 single segment selective, and 9 of 10 multisegment patients received max 50mg dose of doxorubicin. Dose-normalized concentrations reported for all.
  Same distributions apply to doxorubicinol results. In addition, for 1 lobar patient and 8 selective patients, doxorubicinol concentrations were below limit of quantification.
Measure: Mean (Standard Deviation); unit: ng/mL/mg
Arm/Group | Superselective cTACE Doxorubicin (One Segment) | Superselective cTACE (2+ Segments) | Whole Liver Lobe cTACE Doxorubicin
Number analyzed (Participants) | 10 | 10 | 10
ng/mL/mg
  Doxorubicin Cmax normalized dose | 2.67 (2.02) | 3.68 (4.20) | 7.11 (4.24)
  Doxorubicinol Cmax normalized for dose | 0.08 (0.11) | 0.20 (0.22) | 0.34 (0.15)
Statistical Analysis 1: Comparison: Superselective cTACE Doxorubicin (One Segment) vs Superselective cTACE (2+ Segments) vs Whole Liver Lobe cTACE Doxorubicin; To achieve high probability (80% power) to detect 50% change with 5% significance level, calculated total sample size was 30 participants for dose normalized doxorubicin; Test type: Other; p = .036, Kruskal-Wallis — Two-sided p-values <0.05 considered statistically significant
Statistical Analysis 2: Comparison: Superselective cTACE Doxorubicin (One Segment) vs Superselective cTACE (2+ Segments) vs Whole Liver Lobe cTACE Doxorubicin; To achieve high probability (80% power) to detect 50% change with 5% significance level, calculated total sample size was 30 participants for dose normalized doxorubicinol; Test type: Other; p = 0.002, Kruskal-Wallis — Two-sided p-values <0.05 considered statistically significant

2. Primary Outcome: Pharmacokinetics Profile-- Peak of Plasma Concentration
Description: Peak of plasma concentration (Cmax) of doxorubicin and doxorubicinol reported for 10 lobar subjects, 10 superselective subjects with Lipiodol distribution to 1 segment, and 10 superselective subjects with Lipiodol distribution to multiple segments.
Time Frame: 0, 5, 10, 20, 40 minutes, 1, 2, 4, 24 hours, and 3-4 weeks post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Superselective cTACE Doxorubicin (One Segment) | Superselective cTACE (2+ Segments) | Whole Liver Lobe cTACE Doxorubicin
Number analyzed (Participants) | 10 | 10 | 10
ng/mL
  Doxorubicin Cmax | 83.94 (75.09) | 139.66 (117.73) | 334.35 (215.18)
  Doxorubicinol Cmax | 3.79 (5.52) | 7.71 (6.47) | 15.87 (7.57)

3. Primary Outcome: Pharmacokinetics Profile-- Area Under the Concentration Time Curve (Dose Normalized)
Description: Area under the concentration time curve (AUC) reported for doxorubicin and doxorubicinol reported for 10 lobar subjects, 10 superselective subjects with Lipiodol distribution to 1 segment, and 10 superselective subjects with Lipiodol distribution to multiple segments after dose normalization.
Time Frame: 0, 5, 10, 20, 40 minutes, 1, 2, 4, 24 hours, and 3-4 weeks post dose
Measure: Mean (Standard Deviation); unit: ng*h/mL/mg
Arm/Group | Superselective cTACE Doxorubicin (One Segment) | Superselective cTACE (2+ Segments) | Whole Liver Lobe cTACE Doxorubicin
Number analyzed (Participants) | 10 | 10 | 10
ng*h/mL/mg
  Doxorubicin dose normalized AUC | 2.87 (1.95) | 4.44 (4.00) | 7.10 (5.58)
  Doxorubicinol dose normalized AUC | 0.63 (1.16) | 1.32 (2.10) | 1.91 (2.39)
Statistical Analysis 1: Comparison: Superselective cTACE Doxorubicin (One Segment) vs Superselective cTACE (2+ Segments) vs Whole Liver Lobe cTACE Doxorubicin; To achieve high probability (80% power) to detect 50% change with 5% significance level, calculated total sample size was 30 participants for time-concentration-curves for doxorubicin; Test type: Other; p = 0.023, Kruskal-Wallis — Two-sided p-values <0.05 considered statistically significant
Statistical Analysis 2: Comparison: Superselective cTACE Doxorubicin (One Segment) vs Superselective cTACE (2+ Segments) vs Whole Liver Lobe cTACE Doxorubicin; To achieve high probability (80% power) to detect 50% change with 5% significance level, calculated total sample size was 30 participants for time-concentration-curves for doxorubicinol; Test type: Other; p = 0.041, Kruskal-Wallis — Two-sided p-values <0.05 considered statistically significant

4. Primary Outcome: Pharmacokinetics Profile-- Area Under the Concentration Time Curve
Description: Area under the concentration time curve (AUC) reported for doxorubicin and doxorubicinol reported for 10 lobar subjects, 10 superselective subjects with Lipiodol distribution to 1 segment, and 10 superselective subjects with Lipiodol distribution to multiple segments.
Time Frame: 0, 5, 10, 20, 40 minutes, 1, 2, 4, 24 hours, and 3-4 weeks post dose
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Superselective cTACE Doxorubicin (One Segment) | Superselective cTACE (2+ Segments) | Whole Liver Lobe cTACE Doxorubicin
Number analyzed (Participants) | 10 | 10 | 10
ng*h/mL
  Doxorubicin AUC | 114.79 (109.53) | 195.80 (199.40) | 307.87 (195.69)
  Doxorubicinol AUC | 31.61 (57.78) | 62.27 (105.66) | 79.37 (93.67)

5. Primary Outcome: Pharmacokinetics Profile-- Time of Maximum Concentration
Description: Median time of maximum concentration (Tmax) reported for doxorubicin and doxorubicinol reported for 10 lobar subjects, 10 superselective subjects with Lipiodol distribution to 1 segment, and 10 superselective subjects with Lipiodol distribution to multiple segments.
Time Frame: 0, 5, 10, 20, 40 minutes, 1, 2, 4, 24 hours, and 3-4 weeks post dose
Measure: Median (Full Range); unit: hours
Arm/Group | Superselective cTACE Doxorubicin (One Segment) | Superselective cTACE (2+ Segments) | Whole Liver Lobe cTACE Doxorubicin
Number analyzed (Participants) | 10 | 10 | 10
hours
  Median Tmax doxorubicin | 0.53 [0.12 to 1.72] | 0.60 [0.17 to 1.22] | 0.33 [0.15 to 1.47]
  Median Tmax doxorubicinol | 1.20 [0.37 to 4.27] | 1.10 [0.25 to 4.82] | 0.38 [0.15 to 1.47]

6. Secondary Outcome: Number of Participants With Technical Success of cTACE Procedure.
Description: Feasibility/technical success (yes/no) is measured by ability to administer a therapeutic dose, which is determined clinically.
Time Frame: assessed at baseline (at the time of the cTACE procedure)
Measure: Count of Participants; unit: Participants
Arm/Group | Superselective cTACE Doxorubicin (One Segment) | Superselective cTACE (2+ Segments) | Whole Liver Lobe cTACE Doxorubicin
Number analyzed (Participants) | 10 | 10 | 10
Participants | 10 | 10 | 10

7. Secondary Outcome: Assessment and Frequency of Toxicities (Laboratory and Clinical Adverse Events) According to NCI Common Toxicity Criteria for AE (CTCAE) 5.0.
Description: Adverse events assessed by CTCAE 5.0 and stratified by Lipiodol distribution. 30 patients were reviewed for toxicities.
Time Frame: up to 4 weeks post cTACE
Population: 1 participant in the superselective cTACE (2+ segment) population did not experience any adverse events.
Measure: Number; unit: participants
Arm/Group | Superselective cTACE Doxorubicin (One Segment) | Superselective cTACE (2+ Segments) | Whole Liver Lobe cTACE Doxorubicin
Number analyzed (Participants) | 10 | 10 | 10
participants
  Alkaline phosphatase increased (Grade 1) | 0 | 2 | 1
  Aspartate aminotransferase increased (Grade 1) | 0 | 0 | 2
  Alanine aminotransferase increased (Grade 2) | 0 | 0 | 1
  INR increased (Grade 1) | 0 | 2 | 1
  INR increased (Grade 2) | 0 | 1 | 0
  Blood bilirubin increased (Grade 1) | 2 | 4 | 2
  Blood bilirubin increased (Grade 2) | 1 | 0 | 0
  Hypoalbuminemia (Grade 1) | 3 | 2 | 2
  Hyperglycemia (Grade 1) | 3 | 0 | 2
  Hyperglycemia (Grade 3) | 0 | 0 | 1
  Hyperkalemia (Grade 1) | 1 | 0 | 0
  Hyponatremia (Grade 1) | 1 | 1 | 2
  Hyponatremia (Grade 4) | 0 | 1 | 0
  Anemia (Grade 1) | 2 | 0 | 0
  Anemia (Grade 2) | 0 | 0 | 1
  Platelet count decreased (Grade 1) | 0 | 2 | 0
  Platelet count decreased (Grade 2) | 2 | 0 | 1
  White blood cell decreased (Grade 1) | 1 | 2 | 2
  Lymphocyte count decreased (Grade 1) | 0 | 1 | 0
  Lymphocyte count decreased (Grade 2) | 2 | 2 | 2
  Neutrophil count decreased (Grade 1) | 1 | 0 | 0
  Neutrophil count decreased (Grade 3) | 0 | 0 | 1
  Abdominal pain (Grade 1) | 0 | 0 | 1
  Abdominal pain (Grade 2) | 0 | 1 | 3
  Fatigue (Grade 1) | 1 | 0 | 3
  Fatigue (Grade 2) | 1 | 0 | 1
  Fever (Grade 1) | 1 | 1 | 1
  Nausea (Grade 1) | 0 | 1 | 1
  Nausea (Grade 2) | 1 | 0 | 0
  Alopecia (Grade 1) | 0 | 0 | 1
  Anorexia (Grade 1) | 1 | 2 | 1

ADVERSE EVENTS:
Time Frame: Up to 4 weeks post cTACE
Description: Adverse events determined by regular laboratory tests and clinical visits, reviewed by investigators.
Arm/Group | Superselective cTACE Doxorubicin (One Segment) | Superselective cTACE (2+ Segments) | Whole Liver Lobe cTACE Doxorubicin
All-Cause Mortality (participants affected / at risk) | 1/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10 | 1/10 | 0/10
Other Adverse Events (participants affected / at risk) | 10/10 | 9/10 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Superselective cTACE Doxorubicin (One Segment) (N=10) | Superselective cTACE (2+ Segments) (N=10) | Whole Liver Lobe cTACE Doxorubicin (N=10)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Superselective cTACE Doxorubicin (One Segment) (N=10) | Superselective cTACE (2+ Segments) (N=10) | Whole Liver Lobe cTACE Doxorubicin (N=10)
Alkaline phosphatase increased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Aspartate aminotransferase (Investigations) | 0 (0) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
INR increased (Investigations) | 0 (0) | 3 (3) | 1 (1)
Blood bilirubin increased (Investigations) | 3 (4) | 4 (5) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (4) | 2 (2) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 2 (2) | 2 (2) | 1 (1)
White blood cell decreased (Investigations) | 1 (1) | 2 (2) | 2 (2)
Lymphocyte count decreased (Investigations) | 2 (2) | 3 (3) | 2 (2)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4)
Fatigue (General disorders) | 2 (2) | 0 (0) | 4 (4)
Fever (General disorders) | 1 (1) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-04-20): https://cdn.clinicaltrials.gov/large-docs/81/NCT02753881/Prot_SAP_000.pdf
  • Informed Consent Form (2017-04-20): https://cdn.clinicaltrials.gov/large-docs/81/NCT02753881/ICF_001.pdf